CLINICAL TRIAL: NCT02275325
Title: Assessment of the Preoperative Vestibular Rehabilitation Effectiveness on Balance Control Compensation After Vestibular Schwannoma Surgery
Brief Title: Preoperative Vestibular Rehabilitation Effectiveness After Vestibular Schwannoma Surgery
Acronym: ReveSTAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University of Lorraine (Other)
Responsible Party: Principal Investigator, Cecile PARIETTI-WINKLER, University Professor - Hospital Practitioner, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-A01189-38; 140989B-31 (Other: ANSM)
Record Dates: First submitted 2014-10-17; First posted 2014-10-27 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Vestibular Schwannoma
Keywords: Posture; Unilateral vestibular deafferentation; Medical management; Preoperative vestibular rehabilitation; Neural plasticity
MeSH Terms: conditions — Neuroma, Acoustic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preoperative rehabilitation (Experimental): Patients that have a preoperative vestibular rehabilitation before vestibular schwannoma surgery in addition to the usual postoperative vestibular rehabilitation
  Interventions: Other: Preoperative vestibular rehabilitation
- Usual (No Intervention): Group of patients that solely have a postoperative vestibular rehabilitation after vestibular schwannoma surgery

INTERVENTIONS:
Other: Preoperative vestibular rehabilitation — 12 one-hour sessions with exercises of balance on unstable conditions (foam, tilt of the platform, biofeedback)
  Arms: Preoperative rehabilitation

SUMMARY:
Vestibular schwannoma (VS) is a benign tumour from Schwann cells surrounding the vestibular nerve, which slowly grows within the internal auditory canal and then into the cerebellopontine angle, leading to a gradual vestibular dysfunction. The slowly progressive alteration of vestibular function allows the gradual implementation of central adaptive mechanisms called vestibular compensation. The total unilateral vestibular deafferentation induced by the surgical tumour removal suddenly leads to a decompensation of this previously compensated situation, which explains why most patients report severe vertigo immediately after surgery and which is responsible for perturbations of the postural control (Parietti-Winkler et al., 2006, 2008, 2010, 2011). Recently, Gauchard et al. (2013) suggested that preoperative and regular physical activity would limit the adverse effects of surgical removal on balance control. Also, patients benefited faster and better from the postoperative vestibular rehabilitation.

Thus, preoperative vestibular rehabilitation, including physical and balance exercises, could help to limit postoperative balance disorders and promote postoperative balance compensation. This could lead to a decrease in the duration and cost of the postoperative management and faster improvement of quality of life.

DETAILED DESCRIPTION:
To test this hypothesis, the measured and perceived balance control of the patient and the quality of life will be assessed into two groups: one of two groups will receive preoperative vestibular rehabilitation, carried out by a physiotherapist, and the other not. The assessments will be conducted 45 days and 3 days before surgery, and then 8 days, 30 days, 90 days and 365 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral vestibular schwannoma (stage I to IV according to the Koos classification) with an indication for surgery.
* Patients gave their written informed consent
* Patients are affiliated to the french social welfare

Exclusion Criteria:

* Disorders from the motor and/or somesthetic systems (especially the lower limbs)
* Contraindications to the scheduled functional assessments: ear pathology different from vestibular schwannoma such as cholesteatoma of the middle ear, tympanic membrane perforation, etc.
* Refusal of the surgical procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Acute balance compensation | One week after surgery
  Change in composite equilibrium score from baseline to 8 days after surgery. The baseline corresponds to the day before the preoperative rehabilitation and the composite equilibrium (in %) score is calculated over the six conditions of the Sensory Organization Test (Equitest, Neurocom, USA).
  Comparison between both groups (preoperative rehabilitation vs. usual).

SECONDARY OUTCOMES:
Balance compensation at short term | One month after surgery
  Change in composite equilibrium score from baseline to 30 days after surgery. The baseline corresponds to the day before the preoperative rehabilitation and the composite equilibrium (in %) score is calculated over the six conditions of the Sensory Organization Test (Equitest, Neurocom, USA).
  Comparison between both groups (preoperative rehabilitation vs. usual).
Balance compensation at middle term | Three months after surgery
  Change in composite equilibrium score from baseline to 90 days after surgery. The baseline corresponds to the day before the preoperative rehabilitation and the composite equilibrium (in %) score is calculated over the six conditions of the Sensory Organization Test (Equitest, Neurocom, USA).
  Comparison between both groups (preoperative rehabilitation vs. usual).
Balance compensation at long term | One year after surgery
  Change in composite equilibrium score from baseline to 365 days after surgery. The baseline corresponds to the day before the preoperative rehabilitation and the composite equilibrium (in %) score is calculated over the six conditions of the Sensory Organization Test (Equitest, Neurocom, USA).
  Comparison between both groups (preoperative rehabilitation vs. usual).
Preoperative balance compensation | From baseline to three days before surgery
  Change in composite equilibrium score from baseline to three days before surgery. The baseline corresponds to the day before the preoperative rehabilitation and the composite equilibrium (in %) score is calculated over the six conditions of the Sensory Organization Test (Equitest, Neurocom, USA).
  Comparison between both groups (preoperative rehabilitation vs. usual).
Acute change in self-rated dizziness (measured with the Dizziness Handicap Inventory) | One week after surgery
  Change in self-rated dizziness (measured with the Dizziness Handicap Inventory) from baseline to 8 days after surgery. The baseline corresponds to the day before the preoperative rehabilitation.
  Comparison between both groups (preoperative rehabilitation vs. usual).
Change in self-rated dizziness (measured with the Dizziness Handicap Inventory) at short term | One month after surgery
  Change in self-rated dizziness (measured with the Dizziness Handicap Inventory) from baseline to 30 days after surgery. The baseline corresponds to the day before the preoperative rehabilitation.
  Comparison between both groups (preoperative rehabilitation vs. usual).
Change in self-rated dizziness (measured with the Dizziness Handicap Inventory) at middle term | Three months after surgery
  Change in self-rated dizziness (measured with the Dizziness Handicap Inventory) from baseline to 90 days after surgery. The baseline corresponds to the day before the preoperative rehabilitation.
  Comparison between both groups (preoperative rehabilitation vs. usual).
Change in self-rated dizziness (measured with the Dizziness Handicap Inventory) at long term | One year after surgery
  Change in self-rated dizziness (measured with the Dizziness Handicap Inventory) from baseline to 365 days after surgery. The baseline corresponds to the day before the preoperative rehabilitation.
  Comparison between both groups (preoperative rehabilitation vs. usual).
Acute change in self-rated quality of life (measured with WHOQOL-Bref questionnaire) | One week after surgery
  Change in self-rated quality of life (measured with WHOQOL-Bref questionnaire) from baseline to 8 days after surgery. The baseline corresponds to the day before the preoperative rehabilitation.
  Comparison between both groups (preoperative rehabilitation vs. usual).
Change in self-rated quality of life (measured with WHOQOL-Bref questionnaire) at short term | One month after surgery
  Change in self-rated quality of life (measured with WHOQOL-Bref questionnaire) from baseline to 30 days after surgery. The baseline corresponds to the day before the preoperative rehabilitation.
  Comparison between both groups (preoperative rehabilitation vs. usual).
Change in self-rated quality of life (measured with WHOQOL-Bref questionnaire) at middle term | Three months after surgery
  Change in self-rated quality of life (measured with WHOQOL-Bref questionnaire) from baseline to 90 days after surgery. The baseline corresponds to the day before the preoperative rehabilitation.
  Comparison between both groups (preoperative rehabilitation vs. usual).
Change in self-rated quality of life (measured with WHOQOL-Bref questionnaire) at long term | One year after surgery
  Change in self-rated quality of life (measured with WHOQOL-Bref questionnaire) from baseline to 365 days after surgery. The baseline corresponds to the day before the preoperative rehabilitation.
  Comparison between both groups (preoperative rehabilitation vs. usual).
Acute change in vestibular function | One week after surgery
  Change in vestibular function (measured by means of videonystagmography) from baseline to 8 days after surgery. The baseline corresponds to the day before the preoperative rehabilitation and videonystagmographic tests include both pendular and caloric tests.
  Comparison between both groups (preoperative rehabilitation vs. usual).
Change in vestibular function at short term | One month after surgery
  Change in vestibular function (measured by means of videonystagmography) from baseline to 30 days after surgery. The baseline corresponds to the day before the preoperative rehabilitation and videonystagmographic tests include both pendular and caloric tests.
  Comparison between both groups (preoperative rehabilitation vs. usual).
Change in vestibular function at middle term | Three months after surgery
  Change in vestibular function (measured by means of videonystagmography) from baseline to 90 days after surgery. The baseline corresponds to the day before the preoperative rehabilitation and videonystagmographic tests include both pendular and caloric tests.
  Comparison between both groups (preoperative rehabilitation vs. usual).
Change in vestibular function at long term | One year after surgery
  Change in vestibular function (measured by means of videonystagmography) from baseline to 365 days after surgery. The baseline corresponds to the day before the preoperative rehabilitation and videonystagmographic tests include both pendular and caloric tests.
  Comparison between both groups (preoperative rehabilitation vs. usual).
Preoperative change in vestibular function | From baseline to three days before surgery
  Change in vestibular function (measured by means of videonystagmography) from baseline to three days before surgery. The baseline corresponds to the day before the preoperative rehabilitation and videonystagmographic tests include both pendular and caloric tests.
  Comparison between both groups (preoperative rehabilitation vs. usual).

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Parietti-Winkler, MD, PhD, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- University Hospital of Nancy, Nancy, France